CLINICAL TRIAL: NCT05773885
Title: Home Telerehabilitation Based on Serious Games for Continuity of Care in People With Parkinson's Disease
Brief Title: Telerehabilitation in People With Parkinson's Disease
Acronym: TEMPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 21/30
Record Dates: First submitted 2022-10-03; First posted 2023-03-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; Telerehabilitation; Activities of daily living; Quality of life; Belance; Compliance
MeSH Terms: conditions — Parkinson Disease; Patient Compliance

STUDY DESIGN:
Intervention Model Description: This study is a multicentre, single-blind (evaluator), Randomized Controlled Trial (RCT)
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blind to the study protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (EG) (Experimental): The Experimental Group (EG) will carry out 30 sessions (3-5 days/week, for 6-10 weeks) of motor, speech, and cognitive rehabilitation exercises using the VRRS Tablet home TR system (Khymeia srl, Noventa Padovana, Italy).
  Interventions: Device: VRRS Tablet (Khymeia s.r.l., Noventa Padovana, Italy)
- Control Group (CG) (Active Comparator): The Control Group (CG) will carry out 30 sessions (3-5 days/week, for 6-10 weeks) of conventional rehabilitation treatments (including physiotherapy, occupational therapy, speech therapy, psychotherapy) without the use of any technological devices.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: VRRS Tablet (Khymeia s.r.l., Noventa Padovana, Italy) — The patients will carry out motor, speech, and cognitive rehabilitation exercises using the VRRS Tablet (Khymeia s.r.l., Noventa Padovana, Italy).
  The motor exercises will be performed using inertial sensors for the acquisition and processing of the movement performed by the patient. This data is shown to the patient with visual and auditory feedback in a serious games environment. The exercises will cover the rehabilitation of balance and lower limbs, for example Balance on one leg, March in place, Stand on tiptoe, Squat, etc. The physiotherapists involved in the study will define a protocol of exercises in TR mode customized according to the characteristics and needs of the patient. The exercises in the speech therapy and cognitive domains will be defined by the specialized staff based on the characteristics of the patient.
  The duration of the rehabilitation treatments is 9 hours per week.
  Arms: Experimental Group (EG)
Other: Conventional rehabilitation — The patients will carry out conventional rehabilitation treatments (including physiotherapy, occupational therapy, speech therapy, psychotherapy) without the use of any technological devices.
  The motor exercises will concern the rehabilitation of balance, trunk, and lower limbs and will be performed with a physiotherapist who will customize the treatment based on the characteristics and needs of the patient. The occupational therapy, speech therapy, psychotherapy treatments will be defined by the specialized staff based on the characteristics of the patient.
  The duration of the rehabilitation treatments is 9 hours per week.
  Arms: Control Group (CG)

SUMMARY:
Although TeleRehabilitation (TR) is widely accepted as an appropriate model for the provision of professional health services in the field of physiotherapy, with already established standards, guidelines and policies, there are still few studies in the literature on the use of TR as a rehabilitation tool in people with Parkinson's Disease (PD). Therefore, further studies on the efficacy of TR in the management of motor and non-motor symptoms of PD are needed.

The study TEMPO aims at assessing the efficacy (in terms of autonomy in carrying out the activities of daily life) of a home TR program based on serious games in people with PD compared to conventional day-hospital treatment.

DETAILED DESCRIPTION:
The scientific literature has shown that appropriate exercise can decrease some non-motor symptoms of PD such as fatigue, depression, apathy, and cognitive impairment, and it can positively affect motor performance. However, access to rehabilitation centers is often difficult, with logistic and economic barriers for those not living near a specialized hospital. In recent years, the use of technologies has considerably progressed, and, with the development of telemedicine systems, remote treatments have become a viable option for the management of patients with PD.

The TR has the potential to optimize the timing, intensity, and personalization of rehabilitation intervention and offers the opportunity for a flexible implementation of treatment protocols and the ability to monitor patient progress in real-time. In particular, for patients with neurological degenerative pathologies, who need periodical and tailored rehabilitation for the whole life, the TR has proved feasible and effective. The recent systematic review by Vellata found that the literature on TR in people with PD is limited. The published studies on TR for PD showed that it is feasible and effective in maintaining and/or improving some clinical and non-clinical aspects of PD such as: balance and walking, speech and voice, quality of life, patient satisfaction. However, although TR is widely accepted as an appropriate model for the provision of professional health services in the field of physiotherapy, with already established standards, guidelines and policies, there are still few studies in the literature on the use of TR as a rehabilitation tool in people with Parkinson's disease.

In this context, the efficacy of TR in the management of motor and non-motor symptoms of PD has to be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 80 years;
* diagnosis of Parkinson's Disease according to the "Movement Disorders Society's diagnostic criteria";
* Hoehn & Yahr (H&Y) score between 2 and 3 (ON-state);
* absence of dyskinesias assessed by the MDS-UPDRS with a score to items 4.1 and 4.2 ≤ 2;
* absence of cognitive impairment measured by the MoCA total score ≥ 18;
* stabilized drug treatment;
* have access to the Internet for TR;
* have a caregiver available during rehabilitation sessions in TR;
* have sufficient cognitive and linguistic level to understand and comply with study procedures;
* sign informed consent.

Exclusion Criteria:

* having any cognitive problems or low compliance that prevent using the TR system;
* other neurological pathologies, psychiatric complications or personality disorders;
* musculoskeletal diseases that impair movement;
* presence of dyskinesias assessed by the MDS-UPDRS with a score to items 4.1 and 4.2 > 2;
* presence of cognitive impairment measured by the MoCA total score < 18;
* severe cognitive or linguistic deficits (inability to understand and comply with study procedures);
* presence of blurred or low vision problems;
* hearing and speech impairment affecting participation in the system;
* absence of signature of the informed consent.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - part II | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1) and a follow-up (2 months after the end of the treatment, T2)
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assessed motor experiences of daily living (Range 0-52). A higher score indicated more severe symptoms of PD.

SECONDARY OUTCOMES:
Change in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1) and a follow-up (2 months after the end of the treatment, T2)
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contained 6 questions and were assessed by the examiner (Range 0-24). Part IB contained 7 questions on non-motor experiences of daily living which were completed by the participant (Range 0-28). Part II assessed motor experiences of daily living (Range 0-52). It contained 13 questions completed by the participant. Part III assessed the motor signs of PD and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III (Range 0-236). A higher score indicated more severe symptoms of PD.
Change in the Parkinson's Disease Questionnaire-8 (PDQ-8) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1) and a follow-up (2 months after the end of the treatment, T2)
  The Parkinson's Disease Questionaire-8 is a short-form version, derived from the Parkinson's Disease Questionaire-39. It is a self-administered questionnaire, used to measure the quality of life in People with PD. It consists of 8 questions regarding the subject's disease symptoms, each item ranging from 0 to 4, and the responses consist of 0=Never, 1=Occasionally, 2=Sometimes, 3=Often, and 4=Always or cannot do at all, total score ranging from 0 (never have problems/issues) to 32 (always have problems or cannot do at all).
Change in the Montreal Cognitive Assessment (MoCA) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points.
Change in the Lee Silverman Voice Treatment LOUD assessment (LSVT/LOUD) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  Maximum duration of sustained vocal phonation and variation of maximum fundamental frequency according to the LSVT/LOUD assessment protocol.
Change in the Timed Up and Go test (TUG) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  The TUG test assesses mobility, balance, walking ability, and fall risk in older adults. It is a measure of function with correlates to balance and fall risk. The participant is asked to get up from the chair she/he is sitting in, walk the marked distance of 3 meters and return to her/his seat again. The elapsed time is recorded in seconds.
Change in the Timed Up and Go Dual task test (TUG-D) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  The TUG-D test is a dual-task dynamic measure for identifying individuals who are at risk for falls. It evaluates balance with a simultaneous cognitive and motor task. The cognitive task of the test is serial triple subtraction while the TUG test is a motor task. Balance performance will be recorded in seconds.
Change in the mini-Balance Evaluation Systems Test (mini-BESTest) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  The mini-BESTest is a shortened version of the Balance Evaluation Systems Test. It aims to target and identify 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits. The test was shortened based on factor analysis to include dynamic balance only and to improve clinical utilization. It is 36 items scale that evaluates Balance with total score of 28.
Change in the 10-meter WalkTest (10mWT) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  The 10mWT is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Change in the New Freezing of Gait Questionnaire (NFOG-Q) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1) and a follow-up (2 months after the end of the treatment, T2)
  The New Freezing of Gait Questionnaire (NFOG-Q) is a self-reported questionnaire consisting of 9 items that measure freezing of gait (FOG). The NFOG-Q is the renewed version of the FOG-Q, which originally consisted of 6 items. The total score ranges from 0 to 24, and higher scores denote more severe FOG.
Change in the Activities-specific Balance Confidence scale (ABC) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1) and a follow-up (2 months after the end of the treatment, T2)
  Activities-specific balance confidence (ABC) scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It consists of 16 questions gauging the individual's confidence while doing activities. The items are scored on a 0-100% scale. Items are totalled and then averaged. The higher the average score the higher the confidence with balance and the less likely risk there is for falling.

OTHER OUTCOMES:
Gait analysis (GAIT) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  In a subgroup of subjects. Optical tracking system with reflective markers and force plates for measuring (according to a model used in gait analysis) spatio-temporal parameters, joints kinematics and kinetics (joint moments and foot-soil reaction forces) during a 10-meter-long path.
Posturograghy (POSTURE) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks,T1)
  In a subgroup of subjects. Force plate posturography measurements: centre of pressure displacement and velocity parameters. Data will be collected under 2 different conditions: normal standing with eyes open, normal standing with eyes closed. Postural sway will be measured in the anteroposterior and mediolateral directions.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanaz Pournajaf, DPT, Principal Investigator — IRCCS San Raffaele Roma; Prof. Marco Franceschini, MD, Study Chair — IRCCS San Raffaele Roma
Locations (2):
- Italy (2):
  - San Raffaele Cassino, Cassino, Frosinone
  - IRCCS San Raffaele Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures, including assessment results and relevant demographic data, will be shared in compliance with ethical and legal requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after official publication and upon request.
Access Criteria: Access will be granted upon specific request to the Study Chair, Principal Investigator, Sub-Investigator, or Central Study Contact Person. Researchers must submit a formal proposal outlining the intended use of the data, which will be reviewed for scientific merit and ethical compliance. Approved requests will receive access through a secure data-sharing platform.

REFERENCES:
- [Background] Barbour PJ, Arroyo J, High S, Fichera LB, Staska-Pier MM, McMahon MK. Telehealth for patients with Parkinson's disease: delivering efficient and sustainable long-term care. Hosp Pract (1995). 2016;44(2):92-7. doi: 10.1080/21548331.2016.1166922. PMID 26982525
- [Background] Cikajlo I, Hukic A, Dolinsek I, Zajc D, Vesel M, Krizmanic T, Blazica B, Biasizzo A, Novak F, Peterlin Potisk K. Can telerehabilitation games lead to functional improvement of upper extremities in individuals with Parkinson's disease? Int J Rehabil Res. 2018 Sep;41(3):230-238. doi: 10.1097/MRR.0000000000000291. PMID 29757774
- [Background] Linares-Del Rey M, Vela-Desojo L, Cano-de la Cuerda R. Mobile phone applications in Parkinson's disease: A systematic review. Neurologia (Engl Ed). 2019 Jan-Feb;34(1):38-54. doi: 10.1016/j.nrl.2017.03.006. Epub 2017 May 23. English, Spanish. PMID 28549757
- [Background] Magrinelli F, Picelli A, Tocco P, Federico A, Roncari L, Smania N, Zanette G, Tamburin S. Pathophysiology of Motor Dysfunction in Parkinson's Disease as the Rationale for Drug Treatment and Rehabilitation. Parkinsons Dis. 2016;2016:9832839. doi: 10.1155/2016/9832839. Epub 2016 Jun 6. PMID 27366343
- [Background] Vellata C, Belli S, Balsamo F, Giordano A, Colombo R, Maggioni G. Effectiveness of Telerehabilitation on Motor Impairments, Non-motor Symptoms and Compliance in Patients With Parkinson's Disease: A Systematic Review. Front Neurol. 2021 Aug 26;12:627999. doi: 10.3389/fneur.2021.627999. eCollection 2021. PMID 34512495